CLINICAL TRIAL: NCT07340710
Title: Decreasing Edema With a Novel OCS Solution (DENOVO) Trial
Brief Title: Decreasing Edema With a Novel OCS Solution Trial
Acronym: DENOVO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCS-LUN-021925
Record Dates: First submitted 2025-09-10; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Lung Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- OCS Lung (Experimental)
  Interventions: Device: OCS Lung System
- Static Cold Storage (Active Comparator)
  Interventions: Other: Static Cold Storage

INTERVENTIONS:
Device: OCS Lung System — Donor lungs preserved on OCS Lung System
  Arms: OCS Lung
Other: Static Cold Storage — Donor Lungs preserved on Static Cold Storage
  Arms: Static Cold Storage

SUMMARY:
This is a prospective, multicenter randomized trial of lung transplant recipients transplanted with either a DBD or DCD donor lungs. The DENOVO Trial will enroll a total of 300 patients in the OCS arm and 150 patients in the SCS arm. The primary endpoint will be patient & graft survival and freedom of Primary Graft Dysfunction (PGD) grade 3 within the initial 72 hours post-transplantation.

ELIGIBILITY:
Donor Inclusion/Exclusion Criteria

Inclusion Criteria:

* Donor lungs are deemed clinically acceptable for transplantation after physical examination of the donor lungs in the donor and/or on the back table in the donor operating room.
* Eligible for randomization to OCS or SCS treatment arms.

Exclusion Criteria:

- Severe traumatic donor lung injury with air and/or blood leak (as seen on radiological studies, bronchial examinations or final visual physical assessment in donor's chest or back table).

Recipient Inclusion/Exclusion:

Inclusion Criteria:

* Signed informed consent document and authorization to use and disclose protected health information
* Double lung transplant candidate
* Age ≥ 18 years old

Exclusion:

- Participant in any other interventional clinical or investigational trials/programs that may confound the outcomes of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
30-day patient and graft survival with freedom from PGD3 | 30-days post-transplant
  The primary endpoint is 30-day patient and graft survival with freedom from PGD 3 within the initial 72-hours (T0-T72).

IPD SHARING:
Plan to Share IPD: No